CLINICAL TRIAL: NCT03922685
Title: Control of Postprandial Glycemia: the Roles of Diet and Exercise
Brief Title: Effects of Diet and Exercise on Circadian Glycemia
Acronym: GLYCEMIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Northern Michigan University (Other)
Responsible Party: Principal Investigator, Dr. Katarina Borer, Professor, University of Michigan
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00110793
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Glucose Intolerance
MeSH Terms: conditions — Glucose Intolerance | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The same eight subjects participated in counterbalanced order in:
  (1) sedentary morning trial, (2) exercise morning trial, (3) sedentary evening trial, (4) exercise evening trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Morning sedentary arm (Active Comparator): After arriving at MCRU at 7 h, and having eaten three 25%-carbohydrate meals over the previous 24 h, subjects had an antecubital-vein catheter inserted and consumed their fourth 25%-carbohydrate meal at 7:20 h. Over the next 4 hours, subjects reclined on a bed and had 3-ml blood samples collected at 10-min intervals. After the 11:20 blood sample, subjects were released from MCRU.
  This arm is compared to the other three arms.
  Interventions: Combination Product: Dietary manipulation (25% carbohydrate diet) and behavioral (sedentary)
- Morning exercise arm (Active Comparator): After arriving at MCRU at 7 h, and having eaten three 25%-carbohydrate meals over the previous 24 h, subjects had an antecubital-vein catheter inserted and consumed their fourth 25%-carbohydrate meal at 7:20 h. At 8 h, subjects walked on the treadmill at 50% maximal effort. Between 7:20 and 11:20, 3-ml blood samples were collected at 10-min intervals.After the 11:20 blood sample, subjects were released from MCRU.
  This arm is compared to the other three arms.
  Interventions: Combination Product: Dietary manipulation (25% carbohydrate diet) and behavioral (exercise)
- Evening sedentary arm (Active Comparator): After arriving at MCRU at 19 h, and having eaten three 25%-carbohydrate meals over the previous 24 h, subjects had an antecubital-vein catheter inserted and consumed their fourth 25%-carbohydrate meal at 19:20 h. Over the next 4 hours, subjects reclined on a bed and had 3-ml blood samples collected at 10-min intervals. After the 23:20 blood sample, subjects were released from MCRU.
  This arm is compared to the other three arms.
  Interventions: Combination Product: Dietary manipulation (25% carbohydrate diet) and behavioral (sedentary)
- Evening exercise arm (Active Comparator): After arriving at MCRU at 19 h, and having eaten three 25%-carbohydrate meals over the previous 24 h, subjects had an antecubital-vein catheter inserted and consumed their fourth 25%-carbohydrate meal at 19:20 h. At 8 h, subjects walked on the treadmill at 50% maximal effort. Between 19:20 and 23:20, 3-ml blood samples were collected at 10-min intervals.After the 23:20 blood sample, subjects were released from MCRU.
  This arm is compared to the other three arms.
  Interventions: Combination Product: Dietary manipulation (25% carbohydrate diet) and behavioral (exercise)

INTERVENTIONS:
Combination Product: Dietary manipulation (25% carbohydrate diet) and behavioral (exercise) — The 25% carbohydrate diet consisted of Pulmocare-vanilla liquid, white roll, butter, and string cheese in proportions to achieve 33% of weigh-maintenance diet containing 25% carbohydrate, 20% protein, and 55% fat. Exercise was walking 1 hour on level treadmill at 50% of maximal effort starting 40 minutes after the beginning of the meal
  Arms: Evening exercise arm; Morning exercise arm
Combination Product: Dietary manipulation (25% carbohydrate diet) and behavioral (sedentary) — The 25% carbohydrate diet consisted of Pulmocare-vanilla liquid, white roll, butter, and string cheese in proportions to achieve 33% of weigh-maintenance diet containing 25% carbohydrate, 20% protein, and 55% fat. There was no exercise during this trial.
  Arms: Evening sedentary arm; Morning sedentary arm

SUMMARY:
Specific aims of the study are:

1. to evaluate whether a 24-h exposure to a 25%-carbohydrate diet will reduce postprandial glycemia to the same extent in the evening (19 h) as in the morning (7 h),. and
2. to determine whether one hour of post-meal moderate intensity exercise (at 50% of maximal effort) will further reduce postprandial glycemia.

The outcome measures are: plasma concentrations of glucose, insulin, glucose-dependent-insulinotropic peptide (GIP), leptin, and the ketone body beta-hydroxybutyrate.

DETAILED DESCRIPTION:
The two hypotheses in this study are:

1. A 24-h exposure to a 25%-carbohydrate diet will reduce postprandial glycemia to the same extent in the evening (19 h) as in the morning (7 h), and
2. One hour of moderate-intensity exercise (at 50% of maximal effort) will further reduce postprandial glycemia to the same extent in the evening (19 h) as in the morning (7 h).

Eight postmenopausal subjects (age 58.5 years, BMI 25.6 kg/m2) participated in 4 24-h long crossover trials, two terminating at 7h and the other 2 at 19h. At each circadian time one trial required 60 minutes of moderate-intensity exercise (50% of maximal effort), and the other two involved no exercise.

Three 25%-carbohydrate meals prepared by the Michigan Clinical Research Unit (MCRU) kitchen, were eaten at subjects' home, and the fourth was eaten 20 minutes after subjects' arrival at MCRU at either 19 h or 7 h. Blood was collected from antecubital catheter at 10-minute intervals until 23:20 h or 11:20 h, respectively.Plasma was treated with protease inhibitor to preserve GIP, frozen at -80o C until glucose measurements by glucose oxidase, hormone measurements by chemiluminescence, and ketone measurements by Abbott meter strips.

Exercise intensity was determined before the exercise trials on a treadmill from oxygen consumption (VO2) and carbon dioxide production (VCO2) by subjects walking on a treadmill at 3 mph with the treadmill slope increased by 2% every 3 minutes. Maximal effort was established when respiratory exchange ratio (VCO2/VO2) reached or exceeded 1. The treadmill speed and slope at half maximal effort was used during the one-hour exercise bout which was initiated 40 minutes after the start of the meal.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal
* normal blood glucose
* no cholesterol medication
* age between 50 an 65 years
* overweight but not obese
* BMI between 25 and 30 kg/m2
* weight-stable during past 6 months
* exercise less than 20 minutes three times a week

Exclusion Criteria:

* metabolic disease other than hormonally-corrected hypothyroidism
* musculo-skeletal disability that would preclude exercise
* smoker
* do not meet inclusion criteria

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose concentration | Four hours: 19:20 to 23:20 in the evening trials; 7:20 to 11:20 in the morning trials
  The area under the postprandial glucose curve
Postprandial insulin concentration | Four hours: 19:20 to 23:20 in the evening trials; 7:20 to 11:20 in the morning trials
  The area under the postprandial insulin curve

SECONDARY OUTCOMES:
Postprandial glucose-dependent insulinotropic peptide (GIP) concentration | Four hours: 19:20 to 23:20 in the evening trials; 7:20 to 11:20 in the morning trials
  The area under the postprandial GIP curve
Postprandial beta-hydroxybutyrate concentration | Four hours: 19:20 to 23:20 in the evening trials; 7:20 to 11:20 in the morning trials
  The area under the beta-hydroxybutyrate postprandial curve
Postprandial leptin concentration | Four hours: 19:20 to 23:20 in the evening trials; 7:20 to 11:20 in the morning trials
  The area under the leptin postprandial curve

CONTACTS AND LOCATIONS:
Overall Officials: Katarina T Borer, Ph.D., Principal Investigator — Professor Emerita

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers